CLINICAL TRIAL: NCT02709278
Title: A Clinical Challenge Trial to Evaluate Controlled Human Infection With BCG Administered by the Aerosol Inhaled Route Compared With the Intradermal Route in Healthy, BCG-naïve, UK Adult Volunteers
Brief Title: Aerosol BCG Challenge Trial in Healthy UK Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TB041
Record Dates: First submitted 2016-02-12; First posted 2016-03-16 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
Keywords: BCG; Aerosol; Tuberculosis; Challenge
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group 1A: low dose aerosol BCG SSI (Other): 3 volunteers receiving BCG SSI at a dose of 1 x 10^3 cfu by the aerosol inhaled route, followed by bronchoscopy.
  Interventions: Biological: BCG
- Group 1B: medium dose aerosol BCG SSI (Other): 3 volunteers receiving BCG SSI at a dose of 1 x 10^4 cfu by the aerosol inhaled route, followed by bronchoscopy.
  Interventions: Biological: BCG
- Group 1C: standard dose aerosol BCG SSI (Experimental): 12 volunteers receiving BCG SSI at a dose of 1 x 10^5 cfu by the aerosol inhaled route and intradermal saline placebo, followed by bronchoscopy.
  Interventions: Biological: BCG; Other: Saline placebo
- Group 1D: standard dose intradermal BCG SSI (Experimental): 12 volunteers receiving BCG SSI at a dose of 1 x 10^5 cfu by the intradermal route and aerosol inhaled saline placebo, followed by bronchoscopy and punch biopsy at the intradermal injection site.
  Interventions: Biological: BCG; Other: Saline placebo
- Group 2A: lower than standard dose aerosol BCG Bulgaria (Other): 3 volunteers receiving BCG Bulgaria (InterVax) at a dose of 1 x 10^4 cfu by the aerosol inhaled route, followed by bronchoscopy.
  Interventions: Biological: BCG
- Group 2B: close to the standard dose aerosol BCG Bulgaria (Other): 3 volunteers receiving BCG Bulgaria (InterVax) at a dose of 1 x 10^5 cfu by the aerosol route, followed by bronchoscopy.
  Interventions: Biological: BCG
- Group 2C: higher than standard dose aerosol BCG Bulgaria (Other): 3 volunteers receiving BCG Bulgaria (InterVax) at a dose of 1 x 10^6 cfu by the aerosol inhaled route, followed by bronchoscopy.
  Interventions: Biological: BCG
- Group 2D: close to or higher than standard aerosol BCG (Experimental): 3 volunteers receiving 1 x 10^7 cfu aerosol inhaled BCG Bulgaria (InterVax), followed by bronchoscopy 14 days later
  Interventions: Biological: BCG
- Group 2E: close to or higher than standard intradermal BCG (Experimental): 9 volunteers receiving the optimal dose of aerosol inhaled BCG Bulgaria (InterVax) identified from preliminary results obtained from Groups 2C and 2D, and ID saline placebo, followed by bronchoscopy 14 days later
  Interventions: Other: Saline placebo; Biological: BCG
- Group 2F: 1 log lower than Group 2E (Experimental): 12 volunteers will receive aerosol inhaled saline placebo and intradermal BCG Bulgaria (InterVax), at a dose a log lower than 2E then bronchoscopy and punch biopsy
  Interventions: Other: Saline placebo; Biological: BCG

INTERVENTIONS:
Biological: BCG — BCG SSI (Due to a global shortage of BCG SSI, BCG Bulgaria used in Group 2)
  Arms: Group 1A: low dose aerosol BCG SSI; Group 1B: medium dose aerosol BCG SSI; Group 1C: standard dose aerosol BCG SSI; Group 1D: standard dose intradermal BCG SSI
Other: Saline placebo — Saline placebo
  Arms: Group 1C: standard dose aerosol BCG SSI; Group 1D: standard dose intradermal BCG SSI; Group 2E: close to or higher than standard intradermal BCG; Group 2F: 1 log lower than Group 2E
Biological: BCG — BCG Bulgaria (InterVax)
  Arms: Group 2A: lower than standard dose aerosol BCG Bulgaria; Group 2B: close to the standard dose aerosol BCG Bulgaria; Group 2C: higher than standard dose aerosol BCG Bulgaria; Group 2D: close to or higher than standard aerosol BCG; Group 2E: close to or higher than standard intradermal BCG; Group 2F: 1 log lower than Group 2E

SUMMARY:
TB041 is a clinical challenge trial primarily to evaluate the safety of BCG challenge administered by the aerosol inhaled route in healthy, BCG naive UK adults. The trial will also look to evaluate and compare the amount of BCG recovered from the lungs and from the skin, following challenge by either the aerosol or the intradermal route.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (M.tb) is a pathogen found worldwide that infects humans causing tuberculosis (TB), a transmissible disease resulting in very high mortality and morbidity. It is estimated that a third of the world's population is latently infected with M.tb, and these people carry a 10% lifetime risk of developing active life-threatening disease. In 2013, there were 9 million new cases worldwide and 1.5 million people died of TB. Co-infection with human immunodeficiency virus (HIV) greatly increases risk of TB reactivation and death. TB diagnosis is challenging and drug treatment can be prolonged, harmful, costly and complex. For these reasons an effective vaccine is a global public health priority.

Currently to assess vaccine efficacy against TB there is no reliable alternative to large, randomized controlled trials. These efficacy trials for novel TB vaccines are challenging, time consuming and very costly. For other diseases, such as malaria, challenge studies have been informative. The development of a safe controlled human mycobacterial challenge model which would ultimately be validated against field efficacy studies could greatly facilitate TB vaccine development by being a guide for selecting which candidate TB vaccines to take forwards to large efficacy trials.

TB041 is a clinical challenge trial primarily to evaluate the safety of BCG challenge administered by the aerosol inhaled route in healthy, BCG naive UK adults. The trial will also look to evaluate and compare the amount of BCG recovered from the lungs and from the skin, following challenge by either the aerosol or the intradermal route.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-50 years
* Resident in or near Oxford (CCVTM or OUH) or Birmingham (NIHR-WTCRF) for the = duration of the trial period
* Screening IGRA negative
* Chest radiograph normal
* No relevant findings in medical history or on physical examination
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception (see below) for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register volunteer details with a confidential database (The - Over-volunteering Protection Service) to prevent concurrent entry into clinical studies/trials
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

* Previously resident for more than 12 months concurrently in a tropical climate where significant non-tuberculous mycobacterial exposure is likely
* Participation in another research trial involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the trial period
* Prior vaccination with BCG or any candidate TB vaccine
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial challenge date
* Clinically significant history of skin disorder, allergy, atopy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial agent, sedative drugs, or any local or general anaesthetic agents
* Pregnancy, lactation or intention to become pregnant during trial period Any respiratory disease, including asthma
* Current smoker
* Clinically significant abnormality on screening chest radiograph
* Clinically significant abnormality of spirometry
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Current use of any medication taken through the nasal or inhaled route including cocaine or other recreational drugs
* Clinical, radiological, or laboratory evidence of current active TB disease
* Past treatment for TB disease
* Any clinically significant abnormality of screening blood or urine tests
* Positive HBsAg, HCV or HIV antibodies
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the trial or impair interpretation of the trial data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) | Up to day 168
  Collection of AE data at each visit and via diary card for 28 days after challenge.

SECONDARY OUTCOMES:
Quantification of BCG | At day 14
  Quantification of BCG in bronchoalveolar lavage (BAL) sample and intradermal biopsy sample.

OTHER OUTCOMES:
Identification of cellular markers of immunity | Up to day 168
  Established and exploratory markers of innate, cell mediated and humoral immunity in blood and BAL samples will be used to identify cellular markers of immunity to BCG.
Evaluation of aerosol BCG challenge vs intradermal BCG challenge | Up to day 168
  Laboratory markers of cell mediated and humoral immunity, including ex-vivo ELISpot in blood and intracellular cytokine staining in blood and BAL samples will be used to assess which route of challenge is most effective

CONTACTS AND LOCATIONS:
Overall Officials: Professor Helen McShane, Principal Investigator — University of Oxford; Professor Paul Moss, Principal Investigator — University of Birmingham
Locations (3):
- United Kingdom (3):
  - Centre for Clinical Vaccinology and Tropical Medicine , University of Oxford, Oxford, Oxfordshire
  - Oxford University Hospitals- John Warin Ward, University of Oxford, Oxford, Oxfordshire
  - NIHR Wellcome Trust Clinical Research Facility, University of Birmingham, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Satti I, Marshall JL, Harris SA, Wittenberg R, Tanner R, Lopez Ramon R, Wilkie M, Ramos Lopez F, Riste M, Wright D, Peralta Alvarez MP, Williams N, Morrison H, Stylianou E, Folegatti P, Jenkin D, Vermaak S, Rask L, Cabrera Puig I, Powell Doherty R, Lawrie A, Moss P, Hinks T, Bettinson H, McShane H. Safety of a controlled human infection model of tuberculosis with aerosolised, live-attenuated Mycobacterium bovis BCG versus intradermal BCG in BCG-naive adults in the UK: a dose-escalation, randomised, controlled, phase 1 trial. Lancet Infect Dis. 2024 Aug;24(8):909-921. doi: 10.1016/S1473-3099(24)00143-9. Epub 2024 Apr 12. PMID 38621405